CLINICAL TRIAL: NCT07326813
Title: A Multicenter, Randomized, Double-Blind, Placebo-and Active-Controlled Clinical Study to Evaluate the Efficacy and Safety of D-2570 in the Treatment of Moderate to Severe Plaque Psoriasis.
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of D-2570 in the Treatment of Moderate to Severe Plaque Psoriasis.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2570-302
Record Dates: First submitted 2025-12-12; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Evaluate the efficacy of different doses of D-2570 compared with placebo (Experimental)
  Interventions: Drug: D-2570 Tablet; Drug: Placebo
- Evaluate the efficacy of different doses of D-2570 compared with BMS-98165 (Active Comparator)
  Interventions: Drug: D-2570 Tablet; Drug: BMS-986165 Tablet
- Evaluate the safety of D-2570 treatment at different dosages (Experimental)
  Interventions: Drug: D-2570 Tablet
- Evaluate the pharmacokinetics and pharmacodynamics of D-2570 in patients with plaque psoriasis (Experimental)
  Interventions: Drug: D-2570 Tablet

INTERVENTIONS:
Drug: D-2570 Tablet — D-2570 is a novel inhibitor targeting the TYK2 pseudokinase domain
Drug: BMS-986165 Tablet — BMS-986165 is a novel inhibitor targeting TYK2
  Arms: Evaluate the efficacy of different doses of D-2570 compared with BMS-98165
Drug: Placebo — A placebo refers to a tablet that has no therapeutic effect on medication
  Arms: Evaluate the efficacy of different doses of D-2570 compared with placebo

SUMMARY:
This study is a randomized, double-blind, placebo- and active-controlled multicenter clinical trial involving patients with moderate to severe plaque psoriasis.

Safety and efficacy assessments will be conducted during the scheduled study visits throughout the trial. After completing the respective treatment, all subjects will undergo a safety follow-up. Both the investigators and subjects will remain blinded throughout the entire treatment period.

During the study, subjects are required to provide blood samples for pharmacokinetic (PK) and pharmacodynamic (PD) analyses at the time points specified in the trial protocol.

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily participates in this study after providing fully informed consent, signs a written informed consent form, and agrees to comply with the procedures specified in the study protocol;
* Aged between 18 and 70 years old (inclusive) at the time of signing the informed consent form, regardless of gender;
* The investigator assesses that the subject has plaque psoriasis suitable for systemic therapy, and the condition has been stable for ≥ 6 months before signing the informed consent form;
* At the screening stage and Day 1 (D1) of the treatment period, the Psoriasis Body Surface Area (BSA) is ≥10%, the Physician Global Assessment (PGA) score is ≥ 3 points, and the Psoriasis Area and Severity Index (PASI) score is ≥ 12 points;
* Hematology, Blood chemistry and Urinalysis examination were basically normal;
* Male subjects and female subjects of childbearing potential must agree to abstain from sexual intercourse or adopt effective contraceptive measures from the time of signing the informed consent form (ICF) until 30 days after the last administration of the investigational product.

Exclusion Criteria:

* Suffering from any type of psoriasis including erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, inverse psoriasis, or drug-induced psoriasis;
* Having other skin lesions that may interfere with the assessment of treatment outcomes, such as eczema;
* A history of severe herpes zoster/simplex infection;
* A history of tuberculosis, active tuberculosis, latent tuberculosis, or clinical manifestations suggestive of tuberculosis infection
* Having language barriers, or being unwilling or unable to fully understand and cooperate;
* Being pregnant or lactating women;
* Other circumstances that the investigator deems unsuitable for the subject to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2027-04-12 (Estimated); Study Completion 2027-08-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of different doses of D-2570 compared with placebo in the treatment of patients with moderate to severe plaque psoriasis | Treatment for 16 weeks after enrollment
  Psoriasis Area and Severity Index (PASI)
To evaluate the efficacy of different doses of D-2570 compared with placebo in the treatment of patients with moderate to severe plaque psoriasis | Treatment for 16 weeks after enrollment
  Physician Global Assessment (PGA)
To evaluate the efficacy of different doses of D-2570 compared with placebo in the treatment of patients with moderate to severe plaque psoriasis | Treatment for 16 weeks after enrollment
  Dermatology Life Quality Index (DLQI)

SECONDARY OUTCOMES:
To evaluate the efficacy of different doses of D-2570 compared with BMS-986165 in the treatment of patients with moderate to severe plaque psoriasis | Treatment for 16 weeks after enrollment
  Psoriasis Area and Severity Index (PASI)
To evaluate the efficacy of different doses of D-2570 compared with BMS-986165 in the treatment of patients with moderate to severe plaque psoriasis | Treatment for 16 weeks after enrollment
  Physician Global Assessment (PGA)
To evaluate the efficacy of different doses of D-2570 compared with BMS-986165 in the treatment of patients with moderate to severe plaque psoriasis | Treatment for 16 weeks after enrollment
  Dermatology Life Quality Index (DLQI)
To evaluate the safety of different doses of D-2570 in the treatment of patients with moderate to severe plaque psoriasis | Through study completion, an average of 28 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
To evaluate the safety of different doses of D-2570 in the treatment of patients with moderate to severe plaque psoriasis | Through study completion, an average of 28 weeks
  Vital signs: blood pressure
To evaluate the safety of different doses of D-2570 in the treatment of patients with moderate to severe plaque psoriasis | Through study completion, an average of 28 weeks
  Vital signs: body temperature
To evaluate the safety of different doses of D-2570 in the treatment of patients with moderate to severe plaque psoriasis | Through study completion, an average of 28 weeks
  Vital signs: heart rate
To evaluate the safety of different doses of D-2570 in the treatment of patients with moderate to severe plaque psoriasis | Through study completion, an average of 28 weeks
  Vital signs: respiration
To evaluate the physical examination of different doses of D-2570 in the treatment of patients with moderate to severe plaque psoriasis | Through study completion, an average of 28 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
To evaluate the safety of different doses of D-2570 in the treatment of patients with moderate to severe plaque psoriasis | Through study completion, an average of 28 weeks
  12-lead electrocardiogram (ECG) examination: QT Interval
To evaluate the safety of different doses of D-2570 in the treatment of patients with moderate to severe plaque psoriasis | Through study completion, an average of 28 weeks
  12-lead electrocardiogram (ECG) examination: Heart rate
To evaluate the pharmacokinetic characteristics (PK) of different doses of D-2570 in the treatment of patients with moderate to severe plaque psoriasis | Day1, Day15, Day29, Day57, Day85, Day113
  Blood drug concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No